CLINICAL TRIAL: NCT05402748
Title: Safety and Efficacy of Injection of Human Placenta Mesenchymal Stem Cells Derived Exosomes for Treatment of Complex Anal Fistula
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ahmadi tafti, assistant professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRCT20211212053361N1
Record Dates: First submitted 2022-05-25; First posted 2022-06-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Fistula Perianal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exosome cases (Experimental): The patients whose fistula is treated by exosome (40 patients).
  Interventions: Other: placenta-MSCs derived exosomes
- Controls (Placebo Comparator): The patients whose fistula is treated with conventional treatment plan (40 patients).
  Interventions: Other: placenta-MSCs derived exosomes

INTERVENTIONS:
Other: placenta-MSCs derived exosomes — Exosomes are extracellular vesicles that are 30 to 150 nm in diameter. these vesicles are secreted from various cells. Mesenchymal stem cells exhibit immunomodulatory and anti- inflammatory properties by the use of paracrine effects. Exosomes as a vehicle for signaling, are responsible for a major part of cell to cell signaling. The preclinical animal studies manifested high safety and efficacy for MSC derived exosome treatment on various fistulas and inflammatory bowel disease. In this study we aimed to evaluate the safety and efficacy of Placenta-MSCs derived exosomes in treatment of patients with complex preanal fistula (non-crohn's) in phase I and II of clinical trial.

SUMMARY:
Study aim:

Safety of Human Placenta Mesenchymal Stem Cells Derived Exosomes for treatment of complex Anal Fistula 2.Efficacy of Human Placenta Mesenchymal Stem Cells Derived Exosomes for treatment of refractory Anal Fistula 3.Fistula changes in MRI studies, 12 weeks after treatment 4.Evaluation of quality of life in perianal fistula patient's questionnaire score before and 12 weeks after treatment

Participants/Inclusion and exclusion criteria:

inclusion Criteria : 1.Age between 18-70 years old 2.Occurrence of complex perianal fistula 3.Informed consent Exclusion Criteria: 1.Active inflammatory bowel disease 2.Synchronous perianal abscess 3.Alcohol,narcotic and stimulant consumption 4.Having active Hepatitis B,C,HIV or TB 5.Peregnancy and lactation 6.Uncontrolled diabetes mellitus 7.Evidence of surgical contraindication 8.Psychological disorders and noncooperative patient

Intervention groups:

Human Placenta Mesenchymal Stem Cells Derived Exosomes injected in fistula tract of patients with complex perianal Fistula in 3 weekly episodes and it's safety and efficacy was evaluated.

Design:

this study includes two separate groups of cases and controls each consisting of 40 participants randomly allocated for the phase 2 of clinical trial.

Settings and conduct:

Patients with complex perianal fistula referred to Imam Khomeini hospital, will be included in the study if they contain inclusion criteria. The fistula was evaluated by clinical examination and MRI and patients fill the quality of life questionnaire. Exosome injections are performed weekly for consecutive three weeks. Patients will reexamined and fill the questionnaire and MRI will done 12 weeks later. Recent findings will compare with the initial data. During this period, patients are examine for complications.

Main outcome variables:

Discharge amount; External orifice re-epithelialization ; Inflammation, discharge and abscess larger than 2 cm in MR imaging; Quality of life questionnaire score, Inflammatory markers such as CRP, IL-6, TNF-a, calprotectin

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-70 years old
2. Occurrence of complex perianal fistula
3. Informed consent

Exclusion Criteria:

1. Active inflammatory bowel disease
2. Synchronous perianal abscess
3. Alcohol,narcotic and stimulant consumption
4. Having active Hepatitis B,C,HIV or TB
5. Peregnancy and lactation
6. Uncontrolled diabetes mellitus
7. Evidence of surgical contraindication
8. Psychological disorders and noncooperative patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-12-22 (Estimated); Study Completion 2023-03-22 (Estimated)

PRIMARY OUTCOMES:
Safety of injected exosomes | 3 months
  assessing the adverse outcomes after injection such as acute allergic reactions
clinical Efficacy of injected exosomes | 3 months
  assessing the clinical response to therapy which might demonstrate itself as closure of refractory fistulas
inflammatory markers | 3 months
  assessing inflammatory markers through laboratory workup including CRP, IL-6, TNF-a, calprotectin.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Colorectal Surgery, Department of Surgery, Tehran University of Medical Sciences, Tehran, Iran, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided